CLINICAL TRIAL: NCT06779591
Title: Implementation and Effectiveness of the Medication Adherence "CareAide® App" for People with Cardiometabolic Diseases At an Academic Primary Care Clinic in Malaysia: a Hybrid Implementation-effectiveness Study
Brief Title: Implementation and Effectiveness of "CareAide® App" for People with Cardiometabolic Diseases At a Primary Care Clinic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024724-13968; 2024724-13968 (Other: University Malaya Medical Center, Malaysia)
Record Dates: First submitted 2025-01-01; First posted 2025-01-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Diabetes Mellitus Type 2; Dyslipidemia
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Intervention group participants will receive 24 weeks of free, unlimited access to the CareAide® app.
  The CareAide® app will help the intervention group track their medication, view health statistics, help in remote management, act as a health diary, act as a virtual drug cabinet, access medical record files, educate patients and their families, and foster community among afflicted patients.
  Participants will be assisted by the study coordinator to download the App onto their smartphones and how to navigate the app upon recruitment. They will be asked to use the app to manage their medications for a period of 24 weeks. Participants in the IG will participate in the use of the app for from 0 to 24 weeks while the control group will continue with their usual routine. Assessment of adherence levels and pertinent clinical outcomes is scheduled at the end of 24 weeks of the intervention following the enrolment of participants for both study groups.
  Interventions: Other: CareAide® Medication Adherence Mobile Application
- Control Group (No Intervention): Participants in the control group will continue with their usual routine without being aware of the existence of the app. Assessment of adherence levels and pertinent clinical outcomes is scheduled at the end of 24 weeks of the intervention following the enrolment of participants for both study groups.

INTERVENTIONS:
Other: CareAide® Medication Adherence Mobile Application — CareAide® app is one of the mobile apps in assisting and improving patients' adherence to medications. It is an unique health-tech and insure-tech company with expertise in behavioural science, chronic condition management and technology. The app aims to help patients with chronic conditions live a better everyday life and empower their families and the ecosystem around the patients to drive better outcomes. They have the clinically validated approach to improving adherence. Using behavioural science and smart tech, they improve the day-to-day life of patients, and importantly, empower both patients and health care providers with the digital tools and near real-time insights to proactively manage risks, intervene early to avoid patient emergencies and to help to provide a better customer satisfaction.
  Arms: Intervention Group

SUMMARY:
This study aims to explore the barriers and facilitators to implement CareAide® app among healthcare providers and patients at a primary care clinic in Malaysia.

This is an implementation-qualitative research study meaning researchers will collect data regarding the adoption rate, ease of implementation and adoption, and patient's willingness to use the application. The researchers will also compare the effectiveness of the application as a tool to remind patients to take their medicine, by comparing between a group of participants who use the app and another group of participants who do not use the app.

This study requires participants to use an app, then attend some routine follow-ups and be administered blood tests, followed by an interview to collect their opinions, feelings, and experiences.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Medically diagnosed with either hypertension, type 2 diabetes and dyslipidemia for at least 6 months as listed in electronic health records
* Exhibit a low adherence indicated by Malaysia Medication Adherence Assessment Tool (MyMAAT) scores of <54 scores
* Taking at least one type of medication daily, three medications daily or two medications with multiple dosing intervals prescribed,
* Owns and able to use a smartphone
* Able to read English or Malay

Exclusion Criteria:

* Individuals who are pregnant, already using any adherence apps or diagnosed with any terminal illnesses, visually impaired, disability or mental health related illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reach | Before the start of intervention
  The absolute number, proportion, and representativeness of individuals who are willing to participate in a given initiative, intervention, or program.
  A proxy for reach was used and defined as the percentage of patients who gave informed consent to participate out of all patients approached.
Effectiveness | Before the start of the intervention, and at 24 weeks after the intervention
  The impact of CareAide® app on medication adherence using the Malaysia Medication Adherence Assessment Tool (MyMAAT) score, with 12 points being the minimum score and 60 points being the maximum. Patients are classified as moderate & poor adherence if their score is < 54. Patients have good adherence if their score is ≥ 54.
Effectiveness | Before the start of the intervention, and at 24 weeks after the intervention
  The impact of CareAide® app on hypertension, measured by taking the patient's systolic and diastolic blood pressure in mmHg.
Effectiveness | Before the start of the intervention, and at 24 weeks after the intervention
  The impact of CareAide® app on type 2 diabetes by measuring the patient's fasting blood glucose (mmol/L) and HbA1c (%).
Effectiveness | Before the start of the intervention, and at 24 weeks after the intervention
  The impact of CareAide® app on dyslipidaemia outcomes, measured by taking the patient's total cholesterol (mmol/L), low-density lipoprotein (mmol/L), high density lipoprotein (mmol/L), and triglyceride level (mmol/L).
Adoption | Through study completion, an average of 1 year
  The absolute number, proportion, and representativeness of settings and intervention agents (people who deliver the program) who are willing to initiate a program.
  In the case of this study, adoption is measured by finding out the proportion of doctors that agree to deliver the intervention by calculating the number of doctors participated over the total number of doctors involved.
Implementation | At three months and at 24 weeks after the intervention
  At the setting level, implementation refers to the intervention agents' fidelity to the various elements of an intervention's protocol, including consistency of delivery as intended and the time and cost of the intervention.
  At the individual level, implementation refers to clients' use of the intervention strategies.
  Implementation will be assessed by exploring engagement with key components of the CareAide® app. Engagement will be assessed by looking through the app analytics data to see the frequency of usage of various app key components.
Maintenance | Through study completion, an average of 1 year
  The extent to which a program or policy becomes institutionalized or part of the routine organizational practices and policies.
  At the individual level, maintenance has been defined as the long-term effects of a program on outcomes after 6 or more months after the most recent intervention contact.
  This outcome will measure doctors' and patients' willingness to continue with the app, ease of use, perceived value of each program component, an overall rating of the program, and whether or not they would recommend the app use to others through the means of a self-report section on a questionnaire.
  The System Usability Scale (Brooke, 1986) will also be administered to assess the usability of the App. The scale has a minimum score of 10 and a maximum score of 100. The higher the score, the higher the perceived usability of the CareAide® Medication Adherence Mobile Application.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Petaling Jaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No